CLINICAL TRIAL: NCT07055165
Title: Connect2Care: A Randomized Clinical Trial of a Smartphone-based Application for Prostate Cancer Education and Screenings for African American Men
Brief Title: Connect2Care: Prostate Cancer Education and Screenings for African American Men
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18003
Record Dates: First submitted 2025-06-13; First posted 2025-07-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Health Behavior
MeSH Terms: conditions — Prostatic Neoplasms; Health Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genius app (Experimental): The Prostate Cancer Genius app includes the following components: (1) educational content that is consistent with existing evidence and recommendations for prostate cancer and prostate cancer screening but has been adapted for the African American male population and for adults who read at or below the 8th-grade level; (2) real-time messages about the risks of prostate cancer and the benefits of completing a PSA test, placing a special emphasis on screening considerations for individuals with a family history of prostate cancer and/or lower urinary tract symptoms (measured via the American Urological Association Symptom Score); (3) general trivia that also incorporates quiz questions about prostate cancer and the PSA test; (4) African American-specific testimonials and educational videos; (5) optional counseling by African American prostate cancer survivors; and (6) on-demand, automated ordering of a home-based PSA test.
  Interventions: Behavioral: Prostate Cancer Genius App
- Prevention Taskforce app (Active Comparator): The Prevention Taskforce app provides on-demand access to evidence-based recommendations for prostate cancer for men between 55 and 69 (i.e., it can be accessed as needed).
  Interventions: Behavioral: US Prevention Taskforce App

INTERVENTIONS:
Behavioral: Prostate Cancer Genius App — Participants assigned to use the Prostate Cancer Genius App will receive a combination of (a) scheduled and (b) on-demand content prostate cancer for one month. Scheduled content will be delivered on specific days each week using app notifications. Participants will also receive tailored navigation for ordering a home-based PSA kit, including receiving follow-up information from trained medical professionals about their test results.
  Arms: Genius app
Behavioral: US Prevention Taskforce App — Participants assigned to use the US Prevention Task Force app will download the app from Google Play and will be instructed to use the app for one-month to to become more informed about prostate cancer. They will also be instructed to download a companion app from the Google Play store. This companion app will be used to deliver weekly assessments and order a home-based PSA test kit if the participant chooses to so. Participants assigned to the Prevention Taskforce app will receive a brochure providing details about the purpose of the home-based PSA test.
  Arms: Prevention Taskforce app

SUMMARY:
Prostate cancer is the most diagnosed cancer in African American men and the second-leading cause of cancer-related death. The prostate-specific antigen (PSA) test is an early detection screening tool for prostate cancer, however, knowledge about prostate cancer and screening benefits and risks and uptake of PSA screening remains low among African American men. To address this inequity, this project proposes the use of the Connect2Care App to improve knowledge of prostate cancer, screening benefits, risks and increase readiness to complete a PSA test (e.g., intentions, motivation, confidence, and self-efficacy). The primary goal of this study is to evaluate the efficacy of the Connect2Care App in a 30-day randomized control trial compared to an existing app developed by the U.S. Department of Health & Human Services (Prevention Taskforce App). African American men between the ages of 45 and 69 from Oklahoma (N = 266), who are not up to date with PSA screening according to recommended guidelines, will be randomly assigned 1:1 to receive either app. The app feasibility will be assessed: (1) efficacy, evaluated via post-intervention differences in knowledge of prostate cancer, screening benefits and risks, (2) app engagement and accessibility, measured via self-report validated questionnaires, and (3) app acceptability, explored via semi-structured qualitative interviews. We will explore readiness to complete a PSA test and identify predictors of readiness across both study arms. The successful demonstration of the feasibility of the Connect2Care App among African American men living in Oklahoma will support expanding this intervention to African American men nationwide.

DETAILED DESCRIPTION:
Prostate cancer is the most diagnosed cancer in African American men and the second-leading cause of cancer-related death. The prostate-specific antigen (PSA) test is an early detection screening tool for prostate cancer, however, knowledge about prostate cancer and screening benefits and risks and uptake of PSA screening remains low among African American men. To address this inequity, this project proposes the use of the Connect2Care App to improve knowledge of prostate cancer, screening benefits, risks and increase readiness to complete a PSA test (e.g., intentions, motivation, confidence, and self-efficacy). The primary goal of this study is to evaluate the efficacy of the Connect2Care App in a 30-day randomized control trial compared to an existing app developed by the U.S. Department of Health & Human Services (Prevention Taskforce App). African American men between the ages of 45 and 69 from Oklahoma (N = 266), who are not up to date with PSA screening according to recommended guidelines, will be randomly assigned 1:1 to receive either app. The app feasibility will be assessed: (1) efficacy, evaluated via post-intervention differences in knowledge of prostate cancer, screening benefits and risks, (2) app engagement and accessibility, measured via self-report validated questionnaires, and (3) app acceptability, explored via semi-structured qualitative interviews. We will explore readiness to complete a PSA test and identify predictors of readiness across both study arms. The successful demonstration of the feasibility of the Connect2Care App among African American men living in Oklahoma will support expanding this intervention to African American men nationwide.

A. Specific Aims

The overall objectives of this proposal are to: (1) address two key SDOH (i.e., neighborhood and built environment and access to high-quality preventive care); (2) leverage community and individual levels of influence; and (3) implement a social risk screener and social needs referral process, at both community and individual levels, that mitigates significant barriers to PSA screening and timely follow-up care. Our central hypothesis is that combining a traditional community-engaged research intervention with an innovative smartphone app navigation intervention, while providing access to free PSA screening tests and follow-up care at Stephenson Cancer Center (see Letter of Support), will have a meaningful impact on prostate cancer outcomes among AA men in Oklahoma. This hypothesis has been formulated based on our promising pilot data (see Preliminary Studies). To attain our overall objectives, we will recruit a total of 466 AA men, aged 55-69 and not up to date with PSA screening. As such, the following specific aims are proposed:

Aim 1. Conduct a multimodal community outreach intervention to improve awareness of and access to PSA screening. Approach. The intervention will include (1) a culturally tailored Social Media Campaign, geofenced to counties with the greatest AA prostate cancer incidence. Participants who click on the campaign can order a free at-home PSA test. (2) In-person Community Health Events will provide educational information and access to on-site PSA screening via our mobile screening vans. A total of 200 AA men will be accrued across both outreach methods. Outcomes. Awareness will be measured by the reach and penetration of the interventions and access by the number of completed PSA screening tests.

Aim 2. Determine the efficacy of smartphone intervention on at-home PSA screening rates. Approach. A total of 266 AA men will be randomized to a two-arm RCT for 4 weeks. Intervention arms include US Preventive Services Task Force App (control) vs. Prostate Cancer Genius App (Genius App; intervention). In both arms, participants will receive information about prostate cancer and screening, have access to a free at-home PSA test and free follow-up care, and social needs referrals. Participants in the Genius App will also have access to several culturally tailored, novel features to support at-home PSA screening. Outcomes. Efficacy (primary outcome) is determined by PSA screening rates 30 days post-randomization.

Aim 3. Explore the feasibility and acceptability of a social risk screening tool to connect participants to social needs referral services. Approach. After completing a baseline social risk screener, all participants will receive some form of navigation for social needs referral. Navigation will differ by type and intensity. Participants accrued by community outreach will receive One-Time Navigation via a list of referral resources, tailored to their social needs assessment and geography. Participants enrolled in the smartphone intervention will receive Weekly Navigation, which provides more intensive support via a study navigator and geofenced social needs notifications on their study app. Outcomes. Feasibility will be measured by the percentage of participants who complete a social risk screener, and the percentage connected to a referral service. Acceptability will be assessed via qualitative exit interviews (N=80), stratified by social need (high vs. low).

ELIGIBILITY:
Inclusion Criteria:

* Live in Oklahoma
* Self-identify as Black/African American
* Self-identify as male
* Between ages 45-69
* Not currently diagnosed with prostate cancer

Exclusion Criteria:

* Participants will be excluded if they are not interested in using a phone app for 30 days
* Has taken a PSA test or has completed PSA screening within the past two years

Ages: 45 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 466 (Estimated)
Dates: Start 2025-07-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Awareness | 30 Days
  Awareness will be measured by reach and penetration of the intervention. For the Social Media Campaign, reach will be determined by the percentage of participants who successfully engage with intervention and will be calculated by the number of impressions (i.e., number of times adverts are seen) divided by the number of times participants engaged with the intervention (i.e., click through rate). This will determine a click through rate, which can be calculated per study ad and geographic region. For the Community Health Events, reach will be determined by the number of events hosted and the number of participants who attend. Penetration will also be explored through a geographic informational systems (GIS) analysis to better understand whether spatial (e.g., distance to CHCO sites) and/or participant-level characteristics (e.g., age) were associated with greater likelihood to engage with the intervention (both Social Media Campaign and Community Health Events) and/or complete a PSA.

SECONDARY OUTCOMES:
Access | 30 Days
  Access will be measured by the number of PSA tests completed. The pre- and post-test surveys will assess sociodemographic characteristics, knowledge, attitudes and beliefs about prostate cancer and readiness to screen

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Neil, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- TSET Health Promotion Research Center, Oklahoma City, Oklahoma, United States